CLINICAL TRIAL: NCT06165250
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Co-administrated BR1018B and BR1018C in Patients With Essential Hypertension and Primary Hypercholesterolemia
Brief Title: A Study to Evaluate the Efficacy and Safety of Co-administrated BR1018B and BR1018C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FAEAC-CT-301
Record Dates: First submitted 2023-12-03; First posted 2023-12-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Essential Hypertension; Primary Hypercholesterolemia
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BR1018A-1 + BR1018B + BR1018C (Experimental)
  Interventions: Drug: BR1018A-1; Drug: BR1018B; Drug: BR1018C
- BR1018A + BR1018B-1 + BR1018C (Active Comparator)
  Interventions: Drug: BR1018A; Drug: BR1018B-1; Drug: BR1018C
- BR1018A-1 + BR1018B + BR1018C-1 (Active Comparator)
  Interventions: Drug: BR1018A-1; Drug: BR1018B; Drug: BR1018C-1

INTERVENTIONS:
Drug: BR1018A — One tablet administered alone
  Arms: BR1018A + BR1018B-1 + BR1018C
Drug: BR1018A-1 — One tablet administered alone
  Arms: BR1018A-1 + BR1018B + BR1018C; BR1018A-1 + BR1018B + BR1018C-1
Drug: BR1018B — One tablet administered alone
  Arms: BR1018A-1 + BR1018B + BR1018C; BR1018A-1 + BR1018B + BR1018C-1
Drug: BR1018B-1 — One tablet administered alone
  Arms: BR1018A + BR1018B-1 + BR1018C
Drug: BR1018C — One tablet administered alone
  Arms: BR1018A + BR1018B-1 + BR1018C; BR1018A-1 + BR1018B + BR1018C
Drug: BR1018C-1 — One tablet administered alone
  Arms: BR1018A-1 + BR1018B + BR1018C-1

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of co-administrated BR1018B and BR1018C in patients with essential hypertension and primary hypercholesterolemia

ELIGIBILITY:
<Inclusion Criteria>

Screening Visit (V1)

* Patients with essential hypertension and primary hypercholesterolemia
* If patients are being treated with antihypertensive/antihyperlipidemic drugs at screening, they should be determined to be medically reasonable by investigator about discontinuing existing antihypertensive/antihyperlipidemic drugs during the clinical trial
* Patients under the following criteria at screening:

  * Patients who meet a fasting triglyceride (TG) < 400 mg/dL and LDL-C ≤ 250 mg/dL
  * Patients who meet the following criteria, depending on whether antihypertensive drugs were administered within the last 4 weeks

    1. Naïve : 140 mmHg ≤ MSSBP < 180 mmHg and MSDBP < 110 mmHg
    2. Use antihypertensive drugs : 130 mmHg ≤ MSSBP < 180 mmHg and MSDBP < 110 mmHg

Baseline Visit (V2)

* Patients who meet the following criteria of blood pressure measured in selected reference arm at baseline (According to the clinical situation of each subject, Follow the blood pressure standards(Refer to 2022 The Korean Society of Hypertension Guideline))

  * 140 mmHg(or 130 mmHg) ≤ MSSBP < 180 mmHg
  * MSDBP < 110 mmHg
* Patients who meet fasting serum lipid profile test levels (LDL-C and TG) correspond to cardiovascular risk and risk factors at baseline (Refer to 2022 Korean Guidelines for the Management of Dyslipidemia (the 5th edition))

<Exclusion Criteria>

* Patients with a difference of SiSBP ≥ 20 mmHg and SiDBP ≥ 10 mmHg in blood pressure measured three times on both arms at screening(V1)
* Patients with blood pressure results showing MSSBP ≥ 180 mmHg or MSDBP ≥ 110 mmHg at screening(V1, both arms) and baseline(V2, selected reference arm)
* Patients with a history of secondary hypertension or suspected secondary hypertension; (e.g., coarctation of the aorta, hyperaldosteronism, renal artery stenosis, renal hypertension, pheochromocytoma, Cushing's syndrome and polycystic kidney disease, etc.)
* Patients with a history of secondary hyperlipidemia or suspected hyperlipidemia; (e.g., Chronic renal failure, nephrotic syndrome, dysproteinemia, obstructive liver disease, Cushing's syndrome, hypothyroidism, etc.)
* Patients with hyportensive shock
* Patients with orthostatic hypotension accompanied by symptoms

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Mean sitting systolic blood pressure | 8weeks from Baseline Visit
  The change of mean sitting systolic blood pressure from baseline in BR1018A-1+BR1018B+BR1018C at Week 8 compared to BR1018A+BR1018B-1+BR1018C
LDL-C | 8weeks from Baseline Visit
  The percent of change in LDL-C from baseline in BR1018A-1+BR1018B+BR1018C at Week 8 compared to BR1018A-1+BR1018B+BR1018C-1

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Keimyung University Dongsan Hospital, Daegu
  - Seoul National University Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No